CLINICAL TRIAL: NCT06195007
Title: Motivational Interviewing to Improve Outcomes After Stroke or Transient Ischemic Attack Attributable to Tobacco Use
Brief Title: Motivational Interviewing for Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no research team to conduct study
Sponsor: University of Florida (Other)
Collaborators: Accreditation Council for Graduate Medical Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB202201687
Record Dates: First submitted 2023-12-21; First posted 2024-01-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Acute Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interview (Experimental): Patients included in the study who are being treated by a resident in the MI intervention group will have a motivational interview during their initial hospitalization.
  Interventions: Behavioral: Motivational Interview
- Control (No Intervention): Patients included in the study who are being treated by a resident in the Control group will not have a motivational interview during their hospitalization.

INTERVENTIONS:
Behavioral: Motivational Interview — The motivational interview (MI) is a 10-15 minute patient-centered conversation which will focus on tobacco use. Multiple communication strategies can be employed during the MI, including open-ended questions, affirmative statements, reflective listening, use of a 'confidence ruler', and summarizing. The 'confidence ruler' technique in this patient population involves asking the patient "On a scale of zero to ten, how confident are you that you can stop using tobacco?", and then requesting further information about why they selected a certain number. These communication strategies and techniques are designed to uncover and foster a patient's own internal motivations to change the target behavior.
  Arms: Motivational Interview

SUMMARY:
Motivational interviewing (MI) is a style of communication designed to elicit a person's own reasons for change to drive commitment toward a goal. The goal of this study is to assess the effect of trainee-led MI on patients diagnosed with acute stroke or TIA attributable to modifiable risk factors in comparison to conventional post-stroke counseling, based on patient outcomes, and meaning of work and sense of fulfillment for trainees.

ELIGIBILITY:
Inclusion Criteria:

* Patient presentation consistent with a stroke or TIA
* Patient is a current tobacco user and tobacco use contributed to the stroke
* Resident enrolled in study assigned to Vascular Neurology service during patient admission.

Exclusion Criteria:

* Patient unable or unwilling to follow up in the outpatient stroke clinic after discharge
* Patient has cognitive impairment or aphasia that would preclude meaningful participation in motivational interview (defined as a score of 0 on the National Institute of Health Stroke Scale [NIHSS] questions 1 and 9)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Smoking cessation at 90-day post-discharge follow up | 90 days post-discharge
  Yes or no
Patient rating of ability to improve their health | 90 days post-discharge
  Patient answers question "I am confident that I can work together with my care team to improve my health" with a rating from 1 (do not agree at all) to 10 (completely agree)
Recurrence of stroke / TIA symptoms | 90 days post-discharge
  Yes or no

SECONDARY OUTCOMES:
Patient ability to take stroke prevention medications as prescribed | 90 days post-discharge
  Yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wilson, MD PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No